CLINICAL TRIAL: NCT05070364
Title: Phase 3, Randomized, Open-Label, Parallel Arm Study to Evaluate the Efficacy and Safety of 180 mcg Peginterferon Lambda-1a (Lambda) Subcutaneous Injection for 48 Weeks in Patients With Chronic Hepatitis Delta Virus (HDV) Infection (LIMT-2)
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of Peginterferon Lambda for 48 Weeks in Patients With Chronic HDV
Acronym: LIMT-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIG-LMD-002
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis Delta Virus
Keywords: HDV; Hepatitis D; Viral Hepatitis
MeSH Terms: conditions — Hepatitis D | interventions — peginterferon lambda-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Peginterferon Lambda for 48 weeks (Experimental): Peginterferon Lambda 180 mcg once weekly for 48 weeks with 24 weeks follow-up
  Interventions: Drug: Peginterferon Lambda-1a
- No treatment for 12 weeks (No Intervention): No treatment for 12 weeks followed by Peginterferon Lambda 180 mcg once weekly for 48 weeks and 24 weeks follow-up

INTERVENTIONS:
Drug: Peginterferon Lambda-1a — Immunomodulator
  Other Names: Lambda; Peginterferon Lambda; Pegylated Interferon Lambda
  Arms: Peginterferon Lambda for 48 weeks

SUMMARY:
The Phase 3 LIMT-2 study will evaluate the safety and efficacy of Peginterferon Lambda treatment for 48 weeks with 24 weeks follow-up compared to no treatment for 12 weeks in patients chronically infected with HDV. The primary analysis will compare the proportion of patients with HDV RNA < LLOQ at the 24-week post-treatment visit in the Peginterferon Lambda treatment group vs the proportion of patients with HDV RNA < LLOQ at the Week 12 visit in the no-treatment comparator group.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel arm study that will allocate patients (2:1) with chronic HDV infection to one of two treatment groups: Peginterferon Lambda 180 mcg QW for 48 weeks with 24 weeks follow-up (Arm 1, n=100), or no treatment for 12 weeks followed by Peginterferon Lambda treatment for 48 weeks with 24 weeks of follow-up (Arm 2, n=50). All patients will receive concomitant therapy with a potent 2nd generation anti-HBV nucleos(t)ide analogue (NUC) throughout the study duration.

Data collected during Peginterferon Lambda treatment in Arm 2 will not be included in the primary analysis. The primary purpose of Arm 2 is to provide benchmark data in a parallel reference group for the expected rate of HDV RNA suppression among patients with chronic HDV infection who receive 12 weeks of anti-HBV NUC therapy alone.

Prior to randomization, all patients will enter a run-in phase with 12 weeks of anti-HBV NUC therapy, which will ensure virologic control of HBV (< 100 IU/mL) prior to randomization and start of Peginterferon Lambda therapy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HDV infection documented by a positive HDV antibody test or a positive HDV RNA by RT PCR test for at least 6 months at Screening Visit 2
* Quantifiable HDV RNA by RT-PCR test at Screening Visit 2
* Documented confirmed suppression of HBV DNA (< 100 IU/mL) following at least 12 weeks of anti-HBV NUC treatment with ETV or a TNF-based NUC (TDF or TAF) at Screening Visit 2
* Serum ALT > upper limit of normal (ULN) and < 10 × ULN.
* Patients categorized with Child-Turcotte-Pugh score of ≤ 5 with well compensated liver disease.

Exclusion Criteria:

* History or current evidence of decompensated liver disease (episodes of bleeding esophageal or gastric varices, ascites and/or encephalopathy)
* Treatment with interferons (IFNs) or immunomodulators within 6 months before Screening Visit 2 or refractory to prior IFN treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Durable Virologic Response | 72 weeks
  HDV RNA below the limit of quantitation at 24 weeks post-treatment

CONTACTS AND LOCATIONS:
Locations (48):
- United States (7):
  - Asian Pacific Liver Center at Coalition of Inclusive Medicine, Los Angeles, California
  - Keck Medical Center of USC, Los Angeles, California
  - Stanford Medicine Outpatient Center, Redwood City, California
  - Sutter Pacific Medical Foundation - California Pacific Medical Center, San Francisco, California
  - Rush University Medical Center, Chicago, Illinois
  - NYU Langone Health / NYU Grossman School of Medicine, New York, New York
  - Icahn School of Medicine - Mount Sinai Medical Center, New York, New York
- Belgium (3):
  - University Hospital Antwerp, Edegem, Antwerp
  - CHU Brugmann, Brussels
  - CUB Hôpital Erasme, Brussels
- Bulgaria (2):
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - Medical Center "Nov Rehabilitatsionen Centre" EOOD, Stara Zagora
- France (8):
  - CHU Clermont-Ferrand, Clermont-Ferrand, Clermont-Ferrand Cedex
  - Hopital Saint Eloi, Montpellier, Herault
  - APHP, Hôpital Avicenne, Bobigny
  - Hôpital Beaujon, Clichy
  - Henri-Mondor Hospital, Créteil
  - CHU Grenoble-Alpes, Grenoble
  - CHU de Rouen, Rouen
  - CHU Toulouse, Toulouse
- Georgia (3):
  - LTD,Tbilisi State Medical Univeristy and lngorokva High Medical Technology University Clinic, Tbilisi
  - Infectious diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Academician Nikoloz Kipshidze Central University Clinic, Tbilisi
- Germany (3):
  - ZIM 1, Gastroenterologie, University Hospital Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsmedizin Mainz, I. Med. Klinik, Mainz
- Israel (5):
  - The Liver Diseases Center, Sheba Medical Center, Ramat Gan, Tel Hashomer
  - Emek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
- Italy (3):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Institutul de Cardiologie Chisinau, Chisinau, Moldova
- Romania (4):
  - Dr. Victor Babes Foundation, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - National Institute for Infectious Diseases "Matei Bals", Bucharest
  - Spitalul de Infectioase Galati Romania, Galati
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Turkey (Türkiye) (6):
  - Ankara City Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Ege University Medical Faculty, Bornova
  - Dicle University, Medical Faculty, Diyarbakır
  - Istanbul Universitry-Cerrahapasa, Cerrahpasa School of Medicine, Istanbul
  - Koc University Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No